CLINICAL TRIAL: NCT05103085
Title: Screening for Hepatitis C Using a Rapid Diagnostic Orientation Test (TROD) in Patients Over 50 Years Old in the Digestive Endoscopy Department of the Europeen Hospital Marseille
Acronym: TROCENDO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 21-24
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2021-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Patient undergoing digestive endoscopy and aged 50 years and over
  Interventions: Diagnostic Test: Rapid diagnostic orientation test (TROD) for Hepatitis C

INTERVENTIONS:
Diagnostic Test: Rapid diagnostic orientation test (TROD) for Hepatitis C — Inclusion of patients during the consultation with the gastroenterologist, before hospitalization in the digestive endoscopy department. Each consenting patient benefits from a HCV screening using TROD on the day of their hospitalization in the department.

SUMMARY:
Chronic viral hepatitis C is a public health problem and several management recommendations are available. According to the French High Authority of Health, hepatitis C screening consists of a targeted screening of people at risk of infection by the virus, in particular drug users, people from countries with a high prevalence of the virus or who have received care in those countries, people transfused before 1992, or people who are or have beenincarcerated .

French government recommendations aim to achieve elimination of hepatitis C virus HCV (as early as 2025) and since April 2018 the European Hospital Marseille is engaged in this battle and organizes every year "the day without hepatitis" in the hospital.

Since 2017, direct-acting antiviral treatments have become available in France to all patients infected with HCV, regardless of the degree of severity of their disease. These treatments are effective in more than 95% of cases and, in 2019, 18,000 people were cured. As of today, it is estimated that there are still 110,000 people likely to be treated in France. Among them, 75,000 are unaware of being HCV positive, people who need to be tested.

With one of the largest volumes of digestive endoscopic examinations in France, the European Hospital Marseille may be a significant source of screening for hepatitis C.

Our study proposes to evaluate hepatitis C screening in consenting patients hospitalized in the endoscopy department at the European Hospital Marseille.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 50
* Giving free and informed written consent
* Being affiliated with or benefiting from a social security scheme

Exclusion Criteria:

- Patient unable to express consent

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 50 and over hospitalized in the digestive endoscopy department
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients aged 50 and over tested positive for chronic viral hepatitis C during gastrointestinal endoscopy. | 16 months

SECONDARY OUTCOMES:
Number of patients who refuse viral screening | 16 months
Investigation and identification of potential risk factors in patients diagnosed positive for chronic viral hepatitis C | 16 months
Number of viremic patients without risk factor | 16 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Européen Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No